CLINICAL TRIAL: NCT02905838
Title: Comparison of the Esthetic and Clinical Performance of Implant Supported All Ceramic Crowns Using Two Different Ceramic Abutment Types
Brief Title: Comparison of Two Implant Prosthetic Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abutment Study
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Failure of Dental Prosthesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anatomic e.max Abutment (Active Comparator): Implant-supported single crown was fabricated using a prefabricated stock abutment made of yttrium oxide partially stabilized tetragonal zirconia polycrystalline (Y-TZP) (Anatomic IPS e.max Abutment, straight, color M1, Ivoclar, Liechtenstein) and pressed ceramic (fluorapatite glass-ceramic, IPS e.max ZirPress, Ivoclar, Liechtenstein) using the cut-back technique and hand veneered with a thin layer of fluorapatite veneering ceramic (fluorapatite veneering ceramic, IPS e.max Ceram, Ivoclar, Liechtenstein).
  Interventions: Device: Anatomic e.max Abutment
- CAD/CAM CARES Abutment (Active Comparator): Implant-supported single crown was fabricated using an individualized CAD/CAM abutment made of Y-TZP (CARES® Abutment, Institut Straumann AG, Basel, Switzerland) and hand build-up veneering ceramic technique (fluorapatite veneering ceramic, IPS e.max Ceram, Ivoclar, Liechtenstein).
  Interventions: Device: CAD/CAM CARES Abutment

INTERVENTIONS:
Device: Anatomic e.max Abutment — Implant-supported single crown was fabricated using a prefabricated stock abutment made of yttrium oxide partially stabilized tetragonal zirconia polycrystalline (Y-TZP) (Anatomic IPS e.max Abutment, straight, color M1, Ivoclar, Liechtenstein) and pressed ceramic (fluorapatite glass-ceramic, IPS e.max ZirPress, Ivoclar, Liechtenstein) using the cut-back technique and hand veneered with a thin layer of fluorapatite veneering ceramic (fluorapatite veneering ceramic, IPS e.max Ceram, Ivoclar, Liechtenstein).
  Arms: Anatomic e.max Abutment
Device: CAD/CAM CARES Abutment — Implant-supported single crown was fabricated using an individualized CAD/CAM abutment made of Y-TZP (CARES® Abutment, Institut Straumann AG, Basel, Switzerland) and hand build-up veneering ceramic technique (fluorapatite veneering ceramic, IPS e.max Ceram, Ivoclar, Liechtenstein).
  All implant-supported crowns were fabricated in the same dental laboratory by the same dental technician (Dominique Vinci, Geneva, Switzerland). The implants were placed by experienced oral surgeons in a prosthetic ideal position.
  Arms: CAD/CAM CARES Abutment

SUMMARY:
To assess and compare the esthetic outcome and clinical performance of anterior maxillary all ceramic implant single crowns based either on prefabricated zirconia abutment veneered with pressed ceramics or on a CAD/CAM (computer-aided design and computer-aided manufacturing) CARES® abutment veneered with hand build-up technique.

Participants will be recruited from the patient population who has previously received dental implant treatment, received a provisional restoration and met the inclusion and exclusion criteria according to the study protocol. After final impression, patients will be randomised into Group A (prefabricated anatomic abutments ): one-piece screw retained single crown using a press technique (fluorapatite glass-ceramic, e.max ZirPress) with cut-back technique or Group B (CAD/CAM CARES® abutments): one- piece screw retained single crown with a hand build-up technique (fluorapatite veneering ceramic, e.max Ceram). One week after final restoration (base line visit) the primary and secondary outcome parameters will be assessed. The patients will be followed up to 5 years after final restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have voluntarily signed the informed consent form before any study-related action
2. Males and females with at least 18 years of age
3. Single tooth gaps in the anterior maxilla position 14-24 (FDI)
4. Successfully osseointegrated single tooth implant inserted at least 16 weeks after tooth extraction
5. Full mouth plaque index according to O'Leary ≤ 25%
6. Implant axis compatible with transocclusal screw retention (screw access palatal of incisal edges)

Exclusion Criteria:

1. Systemic disease that would interfere with dental implant therapy
2. Any contraindications for oral surgical procedures
3. History of local irradiation therapy
4. Patients who smoke >10 cigarettes per day or tobacco equivalents or chew tobacco
5. Subjects who had undergone administration of any investigational device within 30 days of enrolment in the study
6. Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance
7. Physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene
8. Pregnant or breastfeeding women
9. Existing implants in the adjacent position
10. Removable dentures or un-restored tooth gaps in the opposing dentition
11. Patients with inadequate oral hygiene or unmotivated for adequate home care
12. Probing pocket depth of ≥ 4 mm on one of the teeth immediately adjacent to the dental implant site
13. Lack of primary stability of the implant
14. Inappropriate implant position for the prosthetic requirements
15. Major simultaneous augmentation procedures
16. Insufficient stability of the implant
17. Screw access position located too close to the planned incisal edge
18. Need of angled abutment due to prosthetic malposition of the implant
19. Height of the abutment is less than 65% of the height of the complete restoration
20. Severe bruxing or clenching habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change in Aesthetic scores: Pink Esthetic Score / White Esthetic Score (PES WES) baseline, 6 months, 1, 3, 5 years performed by 2 independent observers in each center | baseline, 6 months, 1 year, 3 years, 5 years

SECONDARY OUTCOMES:
Change in Clinical Peri-implant Measurements | baseline, 6 months, 1 year, 3 years, 5 years
Implant Success | baseline, 6 months, 1 year, 3 years, 5 years
Survival Rate | baseline, 6 months, 1 year, 3 years, 5 years
Cast Analysis | baseline, 6 months, 1 year, 3 years, 5 years
  Change in reference tooth-crown length and implant-crown length in mm
Number of Technical Complications of the Implant Crown | baseline, 6 months, 1 year, 3 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Julia-Gabriela Wittneben, Dr., Principal Investigator — University of Bern

REFERENCES:
- [Derived] Wittneben JG, Gavric J, Belser UC, Bornstein MM, Joda T, Chappuis V, Sailer I, Bragger U. Esthetic and Clinical Performance of Implant-Supported All-Ceramic Crowns Made with Prefabricated or CAD/CAM Zirconia Abutments: A Randomized, Multicenter Clinical Trial. J Dent Res. 2017 Feb;96(2):163-170. doi: 10.1177/0022034516681767. Epub 2016 Dec 7. PMID 27927884